CLINICAL TRIAL: NCT01129115
Title: Dose Response Study of Exercise for Age-related Cognitive Changes
Brief Title: Dose Response Study of Aerobic Exercise in Older Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jeff Burns, MD (Other)
Responsible Party: Sponsor-Investigator, Jeff Burns, MD, Assistant Professor, Director of the Alzheimer & Memory Center & AD Clinical Research Program, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11883
Record Dates: First submitted 2010-05-18; First posted 2010-05-24 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nonexercise control group (Active Comparator)
  Interventions: Behavioral: Nonexercise control group
- Aerobic Exercise Group 1 (Experimental)
  Interventions: Behavioral: Aerobic Exercise Group 1
- Aerobic Exercise Group 2 (Experimental)
  Interventions: Behavioral: Aerobic Exercise Group 2
- Aerobic Exercise Group 3 (Experimental)
  Interventions: Behavioral: Aerobic Exercise Group 3

INTERVENTIONS:
Behavioral: Nonexercise control group — Participants randomized to the nonexercise control group will be asked to maintain their current level of physical activity during the 26-week active study period. They will perform outcome assessments and receive the same telephone checks as the exercise group at baseline, 26 and 52 weeks. The purpose of including a non-exercise control group is to allow adequate comparisons with the low, medium and high exercise dose groups on changes in cognitive and physiologic outcome measures.
  Arms: Nonexercise control group
Behavioral: Aerobic Exercise Group 1 — The 50% group will perform 75 minutes a week of moderate intensity exercise spread over 3 days.
  Arms: Aerobic Exercise Group 1
Behavioral: Aerobic Exercise Group 2 — The 100% group will perform 150 minutes a week of exercise over 3 - 5 days
  Arms: Aerobic Exercise Group 2
Behavioral: Aerobic Exercise Group 3 — The 150% group will perform 225 minutes a week of exercise over 4 - 5 days.
  Arms: Aerobic Exercise Group 3

SUMMARY:
This is a randomized, 26-week study of supervised exercise assessing three doses of exercise in sedentary individuals 65 years of age and over with age-related cognitive changes. A total of 100 subjects (n=25 in each of four groups) will be randomized to a non-aerobic control group, 75 minutes, 150 minutes, or 225 minutes a week of moderate intensity aerobic exercise spread over 3 to 5 days a week for 26 weeks. These exercise doses represent 50%, 100%, or 150% of the recommended exercise dose. Participants will be directly supervised during all exercise sessions for the first two months after which direct supervision will occur during at least one session a week. This is intended to provide increased flexibility while also maintaining direct contact with the participant to enhance adherence. Aerobic fitness, physical function, and cognition will be assessed at baseline and 26 weeks to examine the dose-response relationships.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 65 years or older
* Underactive or sedentary based on the Telephone Assessment of Physical Activity
* Community dwelling with a caregiver willing to accompany the participant to visits to the screening evaluation. The caregiver must visit with the subject more than five times a week.
* Nondemented: Clinical Dementia Rating (CDR) 0
* Adequate visual and auditory abilities to perform all aspects of the cognitive and functional assessments
* Stable doses of medications for at least 30 days prior to screening.
* Likely to participate in all scheduled evaluations and complete the exercise program over 52 weeks

Exclusion Criteria:

* Dementia
* CDR > 0
* Current clinically significant major psychiatric disorder (e.g., Major Depressive Disorder) according to Diagnostic Statistical Manual (DSM)-IV criteria or Geriatric Depression score of 5 or greater.
* Significant psychiatric symptoms (e.g., hallucinations) that could impair the completion of the study
* Current clinically-significant systemic illness likely to result in deterioration of the patient's condition or affect the patient's safety during the study
* History of clinically-evident stroke
* Clinically-significant infection within the last 30 days
* Myocardial infarction or symptoms of coronary artery disease (e.g., angina) in the last two-years.
* Uncontrolled hypertension within the last 6 months
* History of cancer within the last 5 years (except non-metastatic basal or squamous cell carcinoma)
* History of drug or alcohol abuse as defined by DSM-IV criteria within the last 2 years
* Insulin-dependent diabetes mellitus
* Significant pain or musculoskeletal disorder that would prohibit participation in an exercise program

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-05; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Burns, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Vidoni ED, Perales J, Alshehri M, Giles AM, Siengsukon CF, Burns JM. Aerobic Exercise Sustains Performance of Instrumental Activities of Daily Living in Early-Stage Alzheimer Disease. J Geriatr Phys Ther. 2019 Jul/Sep;42(3):E129-E134. doi: 10.1519/JPT.0000000000000172. PMID 29286983
- [Derived] Vidoni ED, Johnson DK, Morris JK, Van Sciver A, Greer CS, Billinger SA, Donnelly JE, Burns JM. Dose-Response of Aerobic Exercise on Cognition: A Community-Based, Pilot Randomized Controlled Trial. PLoS One. 2015 Jul 9;10(7):e0131647. doi: 10.1371/journal.pone.0131647. eCollection 2015. PMID 26158265

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nonexercise Control Group | Aerobic Exercise Group 1 | Aerobic Exercise Group 2 | Aerobic Exercise Group 3
Started | 25 | 25 | 27 | 24
Completed | 23 | 18 | 21 | 15
Not Completed | 2 | 7 | 6 | 9
Not completed — Adverse Event | 1 | 2 | 3 | 3
Not completed — Withdrawal by Subject | 1 | 3 | 1 | 4
Not completed — Protocol Violation | 0 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Participants were recruited as a convenience sample of volunteers through print and online advertising, community talks, and existing databases of individuals willing to be in research studies Participants had to be at least 65, sedentary or underactive a, and free of cognitive impairment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nonexercise Control Group | Aerobic Exercise Group 1 | Aerobic Exercise Group 2 | Aerobic Exercise Group 3 | Total
Number analyzed (Participants) | 25 | 25 | 27 | 24 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (5.8) | 73.5 (5.9) | 72.5 (5.7) | 73.2 (5.3) | 72.9 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 17 | 16 | 65
  Male | 9 | 9 | 10 | 8 | 36

OUTCOME MEASURES:

1. Secondary Outcome: Verbal Memory
Description: Verbal Memory is a latent derived variable derived estimated mean. The reported latent means for this trial are created from the well-known neuropsychological tests: Logical Memory, Delayed Logical Memory, Selective Reminding Task - Free Recall Total, Boston Naming Test.
  Latent variables cannot be measured directly but are derived from a theory-driven confirmatory factor analysis in a structural equation model framework. The latent scores are centered around a mean of 0 and standardized so each value represents a fraction of the standard deviation. There are no limits to the scores. Positive number indicate improved performance.Negative numbers indicate worsening performance.
Time Frame: 26 weeks
Population: Healthy older adults without measurable cognitive decline who did not meet recommended daily activity levels.
Measure: Mean (Standard Error); unit: units on a standardized scale
Arm/Group | Nonexercise Control Group | Aerobic Exercise Group 1 | Aerobic Exercise Group 2 | Aerobic Exercise Group 3
Number analyzed (Participants) | 23 | 18 | 21 | 15
units on a standardized scale | .52 (.09) | .61 (.09) | .47 (.09) | .32 (.09)

2. Primary Outcome: Visuospatial Processing
Description: Visuospatial Processing is a latent derived variable derived estimated mean.The reported latent means for this trial are created from the well-known neuropsychological tests: Block Design, Stroop Color Reading, Digit Symbol Substitution and Trailmaking Test A.
  Latent variables cannot be measured directly but are derived from a theory-driven confirmatory factor analysis in a structural equation model framework. The latent scores are centered around a mean of 0 and standardized so each value represents a fraction of the standard deviation. There are no limits to the scores. Positive number indicate improved performance. Negative numbers indicate worsening performance.
Time Frame: 26 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nonexercise Control Group | Aerobic Exercise Group 1 | Aerobic Exercise Group 2 | Aerobic Exercise Group 3
Number analyzed (Participants) | 23 | 18 | 21 | 15
units on a scale | -.02 (.03) | .19 (.03) | .08 (.03) | .29 (.03)

3. Secondary Outcome: Simple Attention
Description: Simple Attention is a latent derived variable derived estimated mean. The reported latent means for this trial are created from the well-known neuropsychological tests: Digit span Forward and Backward, Letter Numbers Sequencing.
  Latent variables cannot be measured directly but are derived from a theory-driven confirmatory factor analysis in a structural equation model framework. The latent scores are centered around a mean of 0 and standardized so each value represents a fraction of the standard deviation. There are no limits to the scores. Positive number indicate improved performance. Negative numbers indicate worsening performance.
Time Frame: 26 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nonexercise Control Group | Aerobic Exercise Group 1 | Aerobic Exercise Group 2 | Aerobic Exercise Group 3
Number analyzed (Participants) | 23 | 18 | 21 | 15
units on a scale | -.06 (.09) | .11 (.09) | .09 (.09) | .14 (.09)

4. Secondary Outcome: Set Maintenance & Shifting
Description: Set Maintenance and Switching is a latent derived variable derived estimated mean. The reported latent means for this trial are created from the well-known neuropsychological tests: DKEFS Card Sort, Animal and Vegetable Category Fluency.
  Latent variables cannot be measured directly but are derived from a theory-driven confirmatory factor analysis in a structural equation model framework. The latent scores are centered around a mean of 0 and standardized so each value represents a fraction of the standard deviation. There are no limits to the scores. Positive number indicate improved performance. Negative numbers indicate worsening performance.
Time Frame: 26 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nonexercise Control Group | Aerobic Exercise Group 1 | Aerobic Exercise Group 2 | Aerobic Exercise Group 3
Number analyzed (Participants) | 23 | 18 | 21 | 15
units on a scale | .07 (.32) | -.08 (.32) | .14 (.32) | -.13 (.32)

5. Secondary Outcome: Reasoning
Description: Reasoning is a latent derived variable derived estimated mean. The reported latent means for this trial are created from the well-known neuropsychological tests:Letter and Word Inductive Reasoning, Matrix Reasoning.
  Latent variables cannot be measured directly but are derived from a theory-driven confirmatory factor analysis in a structural equation model framework. The latent scores are centered around a mean of 0 and standardized so each value represents a fraction of the standard deviation. There are no limits to the scores. Positive number indicate improved performance. Negative numbers indicate worsening performance.
Time Frame: 26 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nonexercise Control Group | Aerobic Exercise Group 1 | Aerobic Exercise Group 2 | Aerobic Exercise Group 3
Number analyzed (Participants) | 23 | 18 | 21 | 15
units on a scale | .24 (.12) | .08 (.12) | .12 (.12) | .21 (.12)

6. Primary Outcome: Change in Maximal Oxygen Consumption
Description: Maximal Oxygen consumption (VO2 max) is the standard, quantitative measure of aerobic fitness. The physiologic range of scores is approximately 3.5 milliliters of oxygen per kilogram of body weight per minute (ml/kg/min) to approximately 90 (ml/kg/min). Higher numbers indicate greater fitness and positive change indicates increasing fitness. Lower number indicate worse fitness
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Nonexercise Control Group | Aerobic Exercise Group 1 | Aerobic Exercise Group 2 | Aerobic Exercise Group 3
Number analyzed (Participants) | 25 | 25 | 27 | 24
ml/kg/min | -1 (1.6) | 1.4 (1.5) | 1.7 (1.4) | 2.0 (1.9)

7. Primary Outcome: Change in Physical Performance Test
Description: The Physical Performance Test is a 9-item measure of physical function. The range of scores is 0-34. Higher numbers indicate better physical function. Positive change indicates improving function. Negative change indicates decreasing function.
Time Frame: 26 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nonexercise Control Group | Aerobic Exercise Group 1 | Aerobic Exercise Group 2 | Aerobic Exercise Group 3
Number analyzed (Participants) | 25 | 25 | 27 | 24
units on a scale | .2 (1.7) | .1 (2.0) | -.9 (1.9) | .5 (2.3)

ADVERSE EVENTS:
Arm/Group | Nonexercise Control Group | Aerobic Exercise Group 1 | Aerobic Exercise Group 2 | Aerobic Exercise Group 3
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/27 | 0/24
Other Adverse Events (participants affected / at risk) | 2/25 | 8/25 | 16/27 | 15/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nonexercise Control Group (N=25) | Aerobic Exercise Group 1 (N=25) | Aerobic Exercise Group 2 (N=27) | Aerobic Exercise Group 3 (N=24)
Musculoskeletal Soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (8) | 14 (31) | 13 (27) — Musculoskeletal Soreness attributed to exercise
Cardiac (Cardiac disorders) | 1 (1) | 3 (4) | 6 (7) | 6 (7) — Irregular heart rate, angina or EKG change typically seen during cardiopulmonary testing. Events may have been discovered at baseline screening and not attributable to intervention
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) — Coughing or upper respiratory infection made worse by exercise
Infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) — Other infection considered to be exacerbated by exercise

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No